CLINICAL TRIAL: NCT00181532
Title: A Multicentre Randomised Double Blind Placebo-Controlled Phase II Study of Celecoxib and Concurrent Radiotherapy in Stage II-III NSCLC. An Evaluation of Both Tumor Radiosensitization and Normal Tissue Protection
Brief Title: Phase II Study of Celecoxib and Concurrent Radiotherapy in Stage II-III NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02.1376L; CKTO 2003-07; IKL 2003-02; MEC MAASTRO 0205
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: NSCLC; cox-2-inhibitor; radiosensitizer; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
The purpose of this study is to investigate the effect of the adminstration of celecoxib, a cox2-inhibitor in patients with stage II-III non small cell lung cancer receiving radical radiotherapy.

The hypothesis is that celecoxib will increase the remission rate of radiotherapy.

DETAILED DESCRIPTION:
Treatment of non-small cell lung cancer (NSCLC) is difficult, even with the best classical radiation and chemotherapy schedule results remain disappointing. However, there is evidence that increasing the local control rate by delivering radiotherapy either in a short period of time or concomitantly with chemotherapy improves survival. Drawback of a higher radiation dose or addition of chemotherapy is a higher incidence of toxicity. So radiation dose escalation could lead to further improvements of prognosis, but the radiation dose is however limited by radiation-induced lung and esophageal damage.

For NSCLC, non-toxic agents who both increase the effectiveness of radiotherapy and decrease radiation induced lung and esophageal damage are needed. The cox-2-inhibitors seem to be suitable for this purpose. In experimental mice tumor models, it was already shown that COX-2-inhibitors both inhibit tumor growth and enhance the radio-response of the tumor. Moreover, anti-inflammatory agents, such asCOX-2-inhibitors, also lowered the incidence of radiation pneumonitis and esophagitis.

In this study the simultaneous favourable effects of COX-2 inhibitors on tumor response and radiation damage in human cancer patients will be investigated.

Patients will be randomised to receive Celecoxib or placebo. All patients will receive the same radiotherapy treatment. Primary outcome measure is tumor response, assessed by a CT-scan of the thorax, three months after radiotherapy.

The tumor response rate of the experimental group will be compared to the tumor response rate of the control group.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven non-small cell lung cancer
* UICC stage II-III
* WHO performance status 0-2
* less than 10% weight loss the last 6 month
* in case of previous chemotherapy, radiotherapy may start after a minimum of 21 days after the last chemotherapy course
* reasonable lung function: FEV1>30% of the predicted value
* no recent(<3month) severe cardiac disease
* no active peptic ulcer disease
* normal serum bilirubin
* normal serum creatinin
* life expectancy more than 6 month
* measurable cancer
* willing and able to comply with the study prescriptions
* able to give written informed consent before patient registration/randomisation
* no previous radiotherapy to the chest

Exclusion Criteria:

* not not small cell histology, e.g. mesothelioma, lymphoma
* mixed pathology, e.g. non small cell plus small cell cancer
* malignant pleural or pericardial effusion
* concurrent chemotherapy with radiation
* recent (<3month) myocardial infarction
* uncontrolled infectious disease
* distant metastases (stage IV)
* patients with active peptic ulceration or gastrointestinal bleeding in the last year
* patients with a past history of adverse reaction to NSAIDs
* renal disease
* chronic use of NSAIDs, COX-2 inhibitors or Aspirin in dosis >120mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2003-05; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
tumor response rate

SECONDARY OUTCOMES:
local progression free survival 9 months after radiotherapy
radiopneumonitis
lung fibrosis,6 month post radiotherapy
acute esophagitis
quality of life
survival after 1 year
survival after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, PHD, Principal Investigator — Maastricht Radiation Oncology (MAASTRO-clinic)
Locations (1):
- Maastircht Radiation Oncology, Heerlen, Limburg, Netherlands